CLINICAL TRIAL: NCT05822869
Title: Early Prone Positioning Monitored by Electrical Impedance Tomography in Patients With Acute Respiratory Distress Syndrome
Brief Title: Early PP Monitored by EIT in Patients With ARDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Rui Wang, Clinical Professor, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-KE-616
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: acute respiratory distress syndrome, prone position, electrical impedance tomography, mechanical ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EIT guided group (Experimental): During prone ventilation, the PEEP level is adjusted based on EIT monitoring.
  Interventions: Procedure: EIT-guided mechanical ventilation strategy
- Lung protective ventilation group (Other): Lung-protective ventilation strategy during prone positioning that continues the supine position.
  Interventions: Procedure: Lung protective ventilation group

INTERVENTIONS:
Procedure: EIT-guided mechanical ventilation strategy — During prone ventilation, the PEEP level is adjusted based on EIT monitoring. The optimal PEEP is the lowest sum of collapse and overdistension percentages
  Arms: EIT guided group
Procedure: Lung protective ventilation group — Lung-protective ventilation strategy during prone positioning that continues the supine position.
  Arms: Lung protective ventilation group

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) is a syndrome characterized by respiratory distress and refractory hypoxemia caused by pulmonary and extra-pulmonary factors. Despite improvements in diagnosis and treatment in recent years, the mortality rate of severe ARDS is still around 40%. The distribution of lung lesions in ARDS patients is significantly gravity-dependent. Even with lung-protective ventilation strategies, tidal volume is concentrated in the ventral lung region, leading to ventilator-associated lung injury. Prone position ventilation can increase ventilation to the dorsal lung tissue and improve the ventilation-perfusion ratio, thus improving oxygenation. During prone position ventilation in ARDS patients, lung-protective ventilation strategies should be maintained, but with different respiratory mechanics from the supine position, requiring adjustment of ventilator parameters. Electrical Impedance Tomography (EIT) technology can be used for bedside monitoring of mechanically ventilated patients, providing real-time feedback on the patient's ventilation status and having great potential for clinical applications. Investigators believes that EIT monitoring during prone position ventilation in ARDS patients can individualize lung-protective ventilation strategies, minimize alveolar overdistension and collapse, improve the weaning success rate of invasive ventilation, and ultimately improve patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old；
2. Meets the diagnostic criteria for ARDS according to the 2012 Berlin definition；
3. Intubation with invasive mechanical ventilation time < 36 hours；
4. PaO2/FiO2 < 150mmHg.

Exclusion Criteria:

1. Contraindication to the prone position;
2. Contraindication to the EIT;
3. Patients have received extracorporeal membrane oxygenation treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day weaning rate from invasive mechanical ventilation | At 28 days of hospitalization.
  After weaning from invasive mechanical ventilation lasting more than 48 hours, continuation with either high-flow nasal cannula (HFNC) or non-invasive ventilation (NIV).

CONTACTS AND LOCATIONS:
Overall Officials: Rui Wang, Dr., Study Director — Beijing Chao-Yang Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Chao-Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Brower RG, Lanken PN, MacIntyre N, Matthay MA, Morris A, Ancukiewicz M, Schoenfeld D, Thompson BT; National Heart, Lung, and Blood Institute ARDS Clinical Trials Network. Higher versus lower positive end-expiratory pressures in patients with the acute respiratory distress syndrome. N Engl J Med. 2004 Jul 22;351(4):327-36. doi: 10.1056/NEJMoa032193. PMID 15269312
- [Background] Borges JB, Hansen T, Larsson A, Hedenstierna G. The "normal" ventilated airspaces suffer the most damaging effects of mechanical ventilation. Intensive Care Med. 2017 Jul;43(7):1057-1058. doi: 10.1007/s00134-017-4708-1. Epub 2017 Feb 15. No abstract available. PMID 28204859
- [Background] Borges JB, Costa EL, Bergquist M, Lucchetta L, Widstrom C, Maripuu E, Suarez-Sipmann F, Larsson A, Amato MB, Hedenstierna G. Lung inflammation persists after 27 hours of protective Acute Respiratory Distress Syndrome Network Strategy and is concentrated in the nondependent lung. Crit Care Med. 2015 May;43(5):e123-32. doi: 10.1097/CCM.0000000000000926. PMID 25746507
- [Background] Terragni PP, Rosboch G, Tealdi A, Corno E, Menaldo E, Davini O, Gandini G, Herrmann P, Mascia L, Quintel M, Slutsky AS, Gattinoni L, Ranieri VM. Tidal hyperinflation during low tidal volume ventilation in acute respiratory distress syndrome. Am J Respir Crit Care Med. 2007 Jan 15;175(2):160-6. doi: 10.1164/rccm.200607-915OC. Epub 2006 Oct 12. PMID 17038660
- [Background] Scholten EL, Beitler JR, Prisk GK, Malhotra A. Treatment of ARDS With Prone Positioning. Chest. 2017 Jan;151(1):215-224. doi: 10.1016/j.chest.2016.06.032. Epub 2016 Jul 8. PMID 27400909
- [Background] Fernandez R, Trenchs X, Klamburg J, Castedo J, Serrano JM, Besso G, Tirapu JP, Santos A, Mas A, Parraga M, Jubert P, Frutos F, Anon JM, Garcia M, Rodriguez F, Yebenes JC, Lopez MJ. Prone positioning in acute respiratory distress syndrome: a multicenter randomized clinical trial. Intensive Care Med. 2008 Aug;34(8):1487-91. doi: 10.1007/s00134-008-1119-3. Epub 2008 Apr 22. PMID 18427774
- [Background] Taccone P, Pesenti A, Latini R, Polli F, Vagginelli F, Mietto C, Caspani L, Raimondi F, Bordone G, Iapichino G, Mancebo J, Guerin C, Ayzac L, Blanch L, Fumagalli R, Tognoni G, Gattinoni L; Prone-Supine II Study Group. Prone positioning in patients with moderate and severe acute respiratory distress syndrome: a randomized controlled trial. JAMA. 2009 Nov 11;302(18):1977-84. doi: 10.1001/jama.2009.1614. PMID 19903918